CLINICAL TRIAL: NCT05521789
Title: Erector Spinae Blocks for Thoracic Surgery
Brief Title: Erector Spinae Block for Thoracic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCR213913
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Neoplasm; Pulmonary Cancer; Thoracic Diseases; Thoracic Cancer; Thoracic Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Thoracic Diseases; Thoracic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care + ESB Thoracic (Experimental): Patients randomized to this group will receive an erector spinae block in addition to the standard of care treatment
  Interventions: Drug: ESB Thoracic
- Standard of Care (No Intervention): Patients randomized to this group will receive standard of care treatment and NO erector spinae block

INTERVENTIONS:
Drug: ESB Thoracic — Erector spinae thoracic block with bupivacaine
  Arms: Standard of Care + ESB Thoracic

SUMMARY:
The aim of this study is to determine if erector spinae injections with bolus infusions with local anesthetic decrease postsurgical pain and opioid consumption in patients undergoing pulmonary resection surgery.

DETAILED DESCRIPTION:
The research hypothesis for the ESB Thoracic study is that erector spinae blocks with boluses of bupivacaine infusions will decrease patients' postsurgical pain, and thereby decrease the amount of narcotic pain medication used. This will be of particular use in patients who have an anticoagulation need and are not able to receive more invasive nerve blocks.To achieve appropriate exposure for pulmonary resection surgery, whether open or video-assisted, patients have surgical incision in the lateral thoracic region, including disruption to the tributaries of the spinal nerves. Due to this dissection, patients frequently experience significant pain post-operatively. Erector spinae blocks with bupivacaine or ropivacaine with bolus infusion therapy have been shown to treat this spinal nerve pain effectively in rib fractures, thoracoscopic surgeries, and breast surgeries. However, there have been no definitive studies evaluating the effectiveness of erector spinae blocks in postoperative pulmonary resection surgery patients.

It is expected that patients with erector spinae blocks (ESB) will have lower pain visual analogue scores (VAS) and lower total opioid consumption. Learning more about the effectiveness of ESB can help in providing adjunct therapy and thereby minimize post-operative opioids, use of which can add further complications in this group of patients through decreased ventilation and increased atelectasis and hypercarbia. As well, current neuraxial local anesthetic therapy involving epidurals and paravertebral blocks require an absence of anticoagulation in the patient; as a fascial plane block, erector spinae blocks can be safely placed in patients on anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary resection
* 18<age<90

Exclusion Criteria:

* pleurodesis
* decortication
* emergent surgery
* local anesthetic allergy
* intraoperative complication (inadvertent hemorrhage or conversion to open surgery)
* bilateral pulmonary resection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure - Pain Score and Pain Medications (6 hours) | At 6 hours postoperatively
  Study team members will record the patients' visual analogue pain score pain score on the scale of 0-10 (pain score 0-10 numerical rating) at 6 hours, as well as pain medications given. In addition, all patients will receive a Pain Diary with which to record the pain scores and medications received/taken. If a patient is discharged prior to the 24 hours, the patient will continue to fill out the Pain Diary at home up to the 24 hour mark. A phone call by a member of the study team within 72 hours of leaving the hospital will be initiated to review the Pain Diary for data collection purposes.
Outcome Measure - Pain Score and Pain Medications (12 hours) | At 12 hours postoperatively
  Study team members will record the patients' visual analogue pain score pain score on the scale of 0-10 (pain score 0-10 numerical rating) at 12 hours, as well as pain medications given. In addition, all patients will receive a Pain Diary with which to record the pain scores and medications received/taken. If a patient is discharged prior to the 24 hours, the patient will continue to fill out the Pain Diary at home up to the 24 hour mark. A phone call by a member of the study team within 72 hours of leaving the hospital will be initiated to review the Pain Diary for data collection purposes.
Outcome Measure - Pain Score and Pain Medications (24 hours) | At 24 hours postoperatively
  Study team members will record the patients' visual analogue pain score pain score on the scale of 0-10 (pain score 0-10 numerical rating) at 24 hours, as well as pain medications given. In addition, all patients will receive a Pain Diary with which to record the pain scores and medications received/taken. If a patient is discharged prior to the 24 hours, the patient will continue to fill out the Pain Diary at home up to the 24 hour mark. A phone call by a member of the study team within 72 hours of leaving the hospital will be initiated to review the Pain Diary for data collection purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No